CLINICAL TRIAL: NCT02586285
Title: A Randomized Controlled Study on the Effect of S-Adenosyl Methionine Treatment on Anti-tumor Recurrence After Curative Resection of Hepatocellular Carcinoma
Brief Title: Effect of S-Adenosyl Methionine Treatment on Recurrence After Curative Resection of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2014-03-015
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: S-Adenosyl Methionine; Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-Adenosyl Methionine Treatment (Active Comparator): Patients will be treated with S-Adenosyl Methionine treatment after curative resection.
  Interventions: Drug: S-Adenosyl Methionine
- Control group (No Intervention): Patients will be treated without S-Adenosyl Methionine treatment after curative resection.

INTERVENTIONS:
Drug: S-Adenosyl Methionine — 500mg-1000mg,iv,qd
  Other Names: H20090408
  Arms: S-Adenosyl Methionine Treatment

SUMMARY:
The aim of this study is to explore the effect of S-Adenosyl Methionine on recurrence after curative resection of Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is now a major health problem. Although the recent advances in treatment of HCC have significantly improved the prognosis of patients with HCC, the overall survival rate is still unsatisfactory; the 5-year survival rate is only 50-70% even after curative treatment such as hepatic resection and percutaneous radiofrequency ablation. One of the reasons for the poor prognosis of HCC is its high rate of recurrence.However,anti-relapse treatment remains a pressing work to do.

In recent years, some study reported that S-Adenosyl Methionine had an impact on promoting apoptosis and inhibiting the growth on breast cancer, colon cancer,gastric cancer and liver cancer in vitro and vivo.

In this study, we aim to examine whether S-Adenosyl Methionine have an effect on improving patients' recurrence after curative resection of Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age
* Patients preoperatively diagnosed of hepatocellular carcinoma according to the criteria of American Association for the Study of Liver Diseases(AASLD)
* Within Milan criteria
* Without or mild liver cirrhosis and the liver function is Child A class.
* Without any other treatments such as TACE、PEI、PRFA before the surgery
* No evidence for extrahepatic metastasis

Exclusion Criteria:

* Patients with macro tumor thrombus or extrahepatic metastasis.
* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction.
* Subjects accepting other trial drugs or participating in other clinical trials.
* Patients refuse to join our trial.
* Female with pregnancy or during the lactation period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time to tumor recurrence | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China